CLINICAL TRIAL: NCT03956121
Title: Effect of Magnesium Sulfate for Fetal Neuroprotection on Fetal Heart Rate in Case of Prematurity
Brief Title: Magnesium Sulfate (MgSO4) and Fetal Heart Rate (FHR) in Case of Prematurity
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PO18050
Record Dates: First submitted 2018-04-09; First posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-04

CONDITIONS: Fetal Neuroprotection
Keywords: Prematurity; magnesium sulfate; fetal heart rate; short-term variability; fetal neuroprotection
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed group: Exposed group( with magnesium sulfate): fetuses aged 24 + 0AW to 32 + 0AW and benefiting from MgSO4 for neuroprotective purposes, with decision of extraction or spontaneous or induced labour
  Interventions: Other: injection of magnesium sulfate
- Control group: Control group (without magnesium sulfate) : fetuses aged 32 + 1SA to 35 + 0SA without MgSO4, with extraction decision or spontaneous or induced labour

INTERVENTIONS:
Other: injection of magnesium sulfate — The intervention consists to perform a study of the usual fetal heart rate with, in addition, comparison analysis of the short-term variability before and after injection of magnesium sulfate in the exposed group. Two successive short-term variability analyzes will be performed in fetuses of the control group.
  Groups: Exposed group

SUMMARY:
Type of study: prospective descriptive monocentric study

Population: 2 groups: -Exposed group: pregnant patient between 24AW+0day and 32AW+0day receiving magnesium sulfate for fetal neuroprotection in the doubt of premature delivery

* Control group: pregnant patient between 32AW+1day and 35AW+0day in the same context not requiring magnesium sulfate due to their gestationnal age.

Criterion(s) of judgment: Appearance of a change in short-term variability after injection of magnesium sulfate in the exposed group compared to the control group.

Schedule: Inclusion from February 20 to August 31, 2018

Expected results and prospects:

The general impression during my semester at the Jeanne de Flandre maternity clinic in Lille was the variability improves after injection of the magnesium sulfate used in the premature infant as a neuroprotective. The investigators would like to proove that the use of magnesium sulfate as neuroprotective in premature fetuses would improve the fetal heart rate by increasing variability.

In the literature there are numerous publications on the effects of magnesium sulfate used as tocolytic (higher doses) in the threats of premature labour, generally showing a variability and number accelerations decreases without increase the number of decelerations. Is this effect is the same as the doses used for fetal neuroprotection?

Expected benefits of the research:

Magnesium sulfate used on premature infants for fetal neuroprotection has an impact on fetal heart rate, including variability and number of accelerations.

DETAILED DESCRIPTION:
Investigation plan:

Exposed group: fetuses aged 24 + 0AW to 32 + 0AW and benefiting from MgSO4 for neuroprotective purposes, with decision of extraction or spontaneous labour or induced labour:

1 FHR + STV before MgSO4 bolus

1. FHR + STV 10 minutes after the start of the MgSO4 bolus

   Control group: fetuses aged 32 + 1SA to 35 + 0SA without MgSO4, with extraction decision or spontaneous labour or induced labour:
2. FHR + STV at 10 minutes interval : 1 STV at the entrance if suspicion premature labour (in the delivery room) then another 10 minutes after; 2 STV at 10 minutes interval if extraction decision.

Statistical Analysis Plan:

Measurement of the STV value difference before / after MgSO4 in the exposed group and the STV value difference between the 2 measurements in the control group and comparison of these differences.

ELIGIBILITY:
Inclusion Criteria:

Exposed group: fetuses aged 24 + 0AW to 32 + 0AW and benefiting from MgSO4 for neuroprotective purposes, with decision of extraction or spontaneous labour or induced labour:

1 FHR + STV before MgSO4 bolus

1. FHR + STV 10 minutes after the start of the MgSO4 bolus

   Control group: fetuses aged 32 + 1SA to 35 + 0SA without MgSO4, with extraction decision or spontaneous labour or induced labour:
2. FHR + STV at 10 minutes interval : 1 STV at the entrance if suspicion premature labour (in the delivery room) then another 10 minutes after; 2 STV at 10 minutes interval if extraction decision.

Choice of the time of realization of the STV = MgSO4 cross almost immediately the placental barrier after its administration.

Exclusion Criteria:

* Term of labour placement or delivery <24AW or > 35AW1day
* Absence of maternal consent
* Absence of realization of magnesium sulfate in the exposed group by maternal contraindication (Heart failure, Maternal heart rhythm disorder, Digitalis treatment, Severe hydro-electrolytic disorders, Renal insufficiency known or oligoanuria, Myasthenia, Maternal or fetal distress requiring a emergency extraction (<30min delay))
* Absence / impossibility of realization of the STV in the exposed or control group.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Exposed group( with magnesium sulfate): fetuses aged 24 + 0AW to 32 + 0AW and benefiting from MgSO4 for neuroprotective purposes, with decision of extraction or spontaneous or induced labour Control group (without magnesium sulfate) : fetuses aged 32 + 1SA to 35 + 0SA without MgSO4, with extraction decision or spontaneous or induced labour
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2018-05-04 (Actual); Primary Completion 2018-09-02 (Actual); Study Completion 2019-03-02 (Actual)

PRIMARY OUTCOMES:
Short term Variability of foetal rythm | day 0
  the short-term variability measure corresponds to the beat-to-beat fluctuation, within periods of 3.75 seconds. it is measured using an Oxford type of monitoring thanks to an algorithm

SECONDARY OUTCOMES:
accelerations and decelerations of foetal rythm | Day 0
  number of accelerations and number of deceleration, within periods of 3.75 seconds. it is measured using an Oxford type of monitoring thanks to an algorithm

CONTACTS AND LOCATIONS:
Locations (1):
- Damien JOLLY, Reims, France